CLINICAL TRIAL: NCT06075121
Title: The Effect of Abdominal Massage on Feeding Intolerance and Blood Sugar Level in Intensive Care Patients with Diabetes and Continuous Enteral Feeding
Brief Title: Enteral Nutrition and Abdominal Massage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amasya University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AmasyaU-EY-208
Record Dates: First submitted 2023-09-27; First posted 2023-10-10 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2023-10

CONDITIONS: Intensive Care Unit Syndrome
Keywords: massage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Abdominal massage group (Experimental): Patients in the massage group will receive an abdominal massage twice a day for 5 days, between 10.00 in the morning and 22.00 in the evening for 15 minutes.
  Interventions: Other: Abdominal massage
- Control group (No Intervention): Routine treatment and care practices in the hospital will continue for 5 days without any additional intervention and the same data will be evaluated at the same time.

INTERVENTIONS:
Other: Abdominal massage — Patients in the massage group will receive an abdominal massage twice a day for 5 days, between 10.00 in the morning and 22.00 in the evening. Enteral nutrition will be interrupted twice a day for 5 days, between 09.30-10.00 in the morning and 21.30-22.00 in the evening, and patients will receive an abdominal massage for 15 minutes.
  Arms: Abdominal massage group

SUMMARY:
This study will be conducted to determine the effect of abominal massage on feeding intolerance and blood sugar levels in intensive care patients who are continuously feeding enterally and have diabetes.

DETAILED DESCRIPTION:
Introduction: Many multiple and challenging problems are encountered in patients followed in intensive care. The most important of these symptoms is nutritional problems. One of the most commonly used methods in the treatment of nutritional problems is enteral nutrition. In addition to its beneficial results, gastrointestinal problems such as abdominal distension, constipation, diarrhea, nausea and vomiting may be encountered in enteral fed individuals in intensive care units. Although different methods are used in the management of complications that may develop in enterally fed patients, abdominal massage, which is one of the non-invasive nursing practices, has been shown to reduce feeding intolerance and balance blood glucose levels.

Purpose: This study will be conducted to determine the effect of abominal massage applied to intensive care patients who are continuously fed enterally and have diabetes, on feeding intolerance and blood sugar levels.

Method: This study will be conducted using a randomized controlled research design. The research sample will consist of 64 patients hospitalized in the intensive care units of a state hospital in Merzifon and who meet the inclusion criteria. Research data will be collected using the clinical status information form, patient parameters monitoring form, and Bristol stool scale. Patients in the massage group will receive an abdominal massage twice a day for 5 days, between 10.00 in the morning and 22.00 in the evening. For the control group, routine treatment and care practices in the hospital will continue without any additional intervention for these 5 days, and the same data will be evaluated at the same time.

Conclusion: It is thought that abdominal massage applied to intensive care patients with diabetes who are continuously fed enterally will reduce feeding intolerance and affect blood sugar levels.

ELIGIBILITY:
Inclusion Criteria:

The age of 18 years and over

Diagnosed with diabetes mellitus

Having just started continuous enteral feeding via nasogastric tube

Glasgow coma scale >3

Patients who do not have a wound in the abdominal area

Patients without current diarrhea, constipation, vomiting, abdominal distension

Patients who gave their consent to participate in the research

Exclusion Criteria:

Patients who had started enteral feeding before starting the study

Patients who received radiotherapy to the abdominal area

Abdominal surgery within the last three months

Patients with ileus

Patients using medications that affect gastrointestinal motility

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2023-06-12 (Actual); Primary Completion 2024-06-22 (Actual); Study Completion 2024-06-22 (Actual)

PRIMARY OUTCOMES:
Gastric residual volume | 5 days
  Gastric residual volume will be done every four hours. GRV measurement will be made 30 minutes after stopping feeding.
Abdominal Distension | 5 days
  Abdominal Distension be evaluated 30 minutes after stopping feeding. Abdominal distention control will be done using the palpation method.
Bristol stool scale scale | 5 days
  This scale is designed to classify an individual's bowel movements into seven separate categories of stool. According to the "Bristol Stool Consistency Scale", Type 1 and Type 2 indicate constipation, Type 3 and Type 4 indicate normal defecation, and Type 5, Type 6 and Type 7 indicate diarrhea.
Blood sugar | 5 days
  Blood glucose levels will be checked four times a day at 10:00-14:00-18:00 and 22:00.

CONTACTS AND LOCATIONS:
Locations (1):
- Amasya U, Amasya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No